CLINICAL TRIAL: NCT07326163
Title: The Effect of Peppermint Oil Aromatherapy on Pain, Functional Capacity and Cost in Fibromyalgia Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bilecik Seyh Edebali Universitesi (Other)
Collaborators: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, Semanur Bilgiç, Research Assistant, Bilecik Seyh Edebali Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Fibromyalgia
Record Dates: First submitted 2025-12-24; First posted 2026-01-08 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Fibromyalgia; Aromatherapy; Cost
Keywords: Aromatherapy; Fibromyalgia; Pain; Functional Capacity; Cost
MeSH Terms: conditions — Fibromyalgia; Pain | interventions — peppermint oil; almond oil; Duloxetine Hydrochloride

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- peppermint oil (Experimental): This group of patients will be introduced to the tender points where chronic pain is detected in fibromyalgia patients, and the areas where these tender points are located will be divided into six regions, which will be identified with the patient. Subsequently, one drop of peppermint oil will be applied transdermally to the inner surface of the patient's forearm, and the application site will be monitored for allergic reactions such as redness or swelling. Patients who do not report any allergic reactions will apply 2 drops of peppermint oil to each area transdermally with their fingertip at 8:00 a.m. and 8:00 p.m. This application will be performed twice daily by the patient for 2 weeks. For areas inaccessible to the patient, a relative/caregiver will apply 2 drops of peppermint oil. The first dose will be administered by the researcher, who will demonstrate the application to the patient. The patient's opinions will be sought and questions answered during the first dose application
  Interventions: Other: Peppermint Oil
- sweet almond oil (Active Comparator): Patients in this group will be introduced to the six sensitive areas where pain is felt, and the locations will be identified with the patient. The patient will apply 2 drops of sweet almond oil to each sensitive area twice daily, at 8:00 a.m. and 8:00 p.m., using their fingertip. This application will be performed twice daily by the patient for 2 weeks. For sensitive areas that the patient cannot access, a family member/caregiver will apply 2 drops of sweet almond oil. The first dose will be administered by the researcher, who will demonstrate the application to the patient. The patient's opinions will be sought and their questions answered during the first dose administration. Sweet almond oil will be provided to patients in dark-coloured glass bottles with droppers and secure caps that open with firm pressure. Patients will be advised to store sweet almond oil at room temperature.
  Interventions: Other: sweet almond oil
- Duloxetine (Other): Patients in this group will receive treatment planned by a rheumatologist. The pharmacological treatment plan will involve administering duloxetine 60 mg once daily for two weeks, a serotonin-noradrenaline reuptake inhibitor effective on descending pain inhibition pathways in fibromyalgia.
  Interventions: Other: Duloxetine

INTERVENTIONS:
Other: Peppermint Oil — This group of patients will be introduced to the tender points where chronic pain is detected in fibromyalgia patients, and the areas where these tender points are located will be divided into six regions, which will be identified with the patient. Subsequently, one drop of peppermint oil will be applied transdermally to the inner surface of the patient's forearm, and the application site will be monitored for allergic reactions such as redness or swelling. Patients who do not report any allergic reactions will apply 2 drops of peppermint oil to each area transdermally with their fingertip at 8:00 a.m. and 8:00 p.m. This application will be performed twice daily by the patient for 2 weeks. For areas inaccessible to the patient, a relative/caregiver will apply 2 drops of peppermint oil. The first dose will be administered by the researcher, who will demonstrate the application to the patient. The patient's opinions will be sought and questions answered during the first dose application
  Arms: peppermint oil
Other: sweet almond oil — Patients in this group will be introduced to the six sensitive areas where pain is felt, and the locations will be identified with the patient. The patient will apply 2 drops of sweet almond oil to each sensitive area twice daily, at 8:00 a.m. and 8:00 p.m., using their fingertip. This application will be performed twice daily by the patient for 2 weeks. For sensitive areas that the patient cannot access, a family member/caregiver will apply 2 drops of sweet almond oil. The first dose will be administered by the researcher, who will demonstrate the application to the patient. The patient's opinions will be sought and their questions answered during the first dose administration. Sweet almond oil will be provided to patients in dark-coloured glass bottles with droppers and secure caps that open with firm pressure. Patients will be advised to store sweet almond oil at room temperature.
  Arms: sweet almond oil
Other: Duloxetine — Patients in this group will receive treatment planned by a rheumatologist. The pharmacological treatment plan will involve administering duloxetine 60 mg once daily for two weeks, a serotonin-noradrenaline reuptake inhibitor effective on descending pain inhibition pathways in fibromyalgia.
  Arms: Duloxetine

SUMMARY:
This study was designed to evaluate the effect of topically applied peppermint oil (Mentha × piperita) on chronic pain and functional capacity experienced by fibromyalgia patients, as well as its cost-effectiveness.

DETAILED DESCRIPTION:
Fibromyalgia is a chronic pain condition characterized by widespread musculoskeletal pain, hyperalgesia, and allodynia, often associated with other symptoms such as fatigue, poor sleep quality, anxiety, and depression. The main symptoms of fibromyalgia include widespread body pain, tender points, muscle stiffness, and joint stiffness, but it is also accompanied by insomnia, fatigue, mood disorders, cognitive dysfunction, anxiety, depression, and difficulty in maintaining daily activities. Fibromyalgia is the third most common musculoskeletal disorder in terms of prevalence after low back pain and osteoarthritis, with prevalence rates ranging from 1.3% to 8.8% depending on the country. Pain can occur at 18 different points on the head, neck, trunk, and extremities, and can increase throughout the day. The presence of chronic and widespread pain leads to fatigue, sleep disorders, depression, anxiety, helplessness, and mental stress, reducing the quality of life for patients. Additionally, these widespread complaints complicate treatment and increase healthcare costs for patients seeking medical help for fibromyalgia. It is estimated that the total healthcare costs for fibromyalgia patients are three times higher than for other individuals. Both pharmacological and non-pharmacological methods are used in the treatment of fibromyalgia, and aromatherapy is among these methods. Considering the analgesic effects and safe usage profile of peppermint oil, its effectiveness in pain management for fibromyalgia patients is being evaluated. This study aims to assess the impact of topically applied peppermint oil on chronic pain and functional capacity experienced by fibromyalgia patients, as well as its cost-effectiveness.

ELIGIBILITY:
Inclusion criteria for the study:

* Diagnosed with fibromyalgia according to the 2010 American College of Rheumatology diagnostic criteria,
* Experiencing chronic pain,
* Volunteers to participate in the study,
* Aged 18 years or older,

Exclusion criteria for the study:

* Those with painful medical conditions other than fibromyalgia (e.g., migraine, diabetic neuropathy, etc.),
* Those with a chronic respiratory system disease (history of asthma or another reactive airway disease),
* Individuals with compromised skin integrity in the application areas,
* Pregnant and/or breastfeeding women,
* Individuals with neurocognitive impairment who are unable to answer the questionnaire,
* Individuals with a known history of allergies,
* Individuals using any topical products during the application period,
* Individuals receiving other complementary treatments for chronic pain management.

Criteria for discontinuing the study:

* Patients who continue their treatment at a different centre after being included in the study,
* Patients who undergo any medication or treatment changes during the study period,
* Patients who are bothered by the scent of the essential oils used (peppermint oil (Mentha × piperita) and sweet almond oil (Prunus amygdalus var. dulcis), or who develop an allergic reaction to essential oils.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale | 2 weeks
  The visual analogue scale is a commonly used pain assessment tool due to its ease of application, reliability, and sensitivity. It consists of a horizontal line measuring 10 cm in length, with the left end labelled 'no pain' and the right end labelled 'severe pain'. The patient is asked to mark the point on this line that best represents their pain intensity, and then the distance between the patient's mark and the left end is measured. This distance, usually measured in millimetres, is interpreted as a 'score'.
The short-form McGill Pain Questionnaire | 2 weeks
  This scale consists of three sections; the first section contains 15 word groups for describing pain. Eleven of these words assess the sensory dimension of pain, while four assess the perceptual dimension. These descriptive words are rated on an intensity scale from 0 to 3 (0 = none, 1 = mild, 2 = moderate, 3 = severe). In the first section of the scale, a total of three pain scores are obtained: sensory pain score, perceptual pain score, and total pain score. The second section contains six word groups ranging from 'no pain' to 'unbearable pain' to determine the severity of the pain. In the third section, the patient's current pain intensity is assessed using a visual analogue scale.
The Revised Fibromyalgia Impact Questionnaire (FIQR) | 2 weeks
  The Fibromyalgia Impact Questionnaire consists of 21 separate questions. All questions are based on an 11-point numerical rating scale ranging from 0 to 10; 10 indicates the worst possible situation, while 0 means no complaint. The questionnaire consists of three subscales: function, overall impact, and symptoms. The function subscale contains 9 questions, the overall impact subscale contains 2 questions, and the symptoms subscale contains 10 questions. The total score obtained from the items related to function (range 0 to 90) is divided by 3, the total score for general impact (range 0 to 20) remains unchanged as it is divided by 1, and the total score for symptoms (range 0 to 100) is divided by 2 for calculation.
Collection of Cost Data from the Perspective of the Reimbursement Agency (Social Security Institution) | 2 weeks
  Costs from the perspective of the reimbursement agency for patients diagnosed with fibromyalgia who receive pharmacological treatment and treatment with aromatherapy oils will be determined through clinical, administrative, and financial records obtained from the hospital's billing, materials management, pharmacy, purchasing, information processing, and statistics departments. Each expense item related to treatments will be classified in detail through detailed invoice breakdowns obtained from the relevant units. Detailed expenditure items related to treatment methods will be expressed through tables.
Collection of Cost Data from the Direct Patient Cost Perspective | 2 weeks
  A questionnaire prepared using the literature will be used to determine costs from the direct patient cost perspective. Using this form, called the direct patient cost questionnaire, expenses such as consultation, aromatherapy oils, medication, transportation, nutrition, bed, accommodation and other items (clothing, cleaning supplies, etc.) will be collected for each patient. Tables showing all expense items will be prepared based on the cost data obtained.

CONTACTS AND LOCATIONS:
Locations (1):
- Bilecik Training and Research Hospital, Bilecik, Bilecik, Turkey (Türkiye)